CLINICAL TRIAL: NCT04789928
Title: Gentamicine-EDTA, a New Anti-biofilm Strategy for the Conservative Treatment of Catheter-related Infections
Brief Title: Conservative Treatment of Catheter - Related Injections With Gentamicine/EDTA
Acronym: CATH-GE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003
Record Dates: First submitted 2021-01-04; First posted 2021-03-10 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-07

CONDITIONS: Patients With Uncomplicated Long-term Central Venous Catheter-related Biofilm-related Infection

STUDY DESIGN:
Intervention Model Description: This is a pilot phase, non-comparative, non-randomized, multicentric study on 35 patients with uncomplicated LTIVC-related BSI and eligible for a conservative treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with uncomplicated LTIVC-related BSI and eligible (Experimental): Patients included in this study will receive daily injection of genta-EDTA-Na2 lock associated with systemic antibiotics.
  Interventions: Drug: Gentamicins-EDTA

INTERVENTIONS:
Drug: Gentamicins-EDTA — Patients included in this study will receive daily injection (up to 10 days) of genta-EDTA-Na2 lock associated with systemic antibiotics.

SUMMARY:
Catheter-related infections are frequent. Treatment without catheter removal is difficult because of the presence of biofilm. The association of gentamicin and EDTA is active in vitro and in vivo against biofilms formed by Gram positive and Gram negative bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 year-old);
* LTIVC in place (TIVAP or single-line tunnelled catheter);
* LTIVC is functional (it is possible to inject an infusate, but also to draw blood from the catheter);
* LTIVC-related bloodstream infection defined by a positive qualitative paired blood culture with a differential time to positivity ≥ 2 hours (meaning that the culture of the blood drawn from the catheter is positive at least 2 hours before the culture of the blood drawn from a peripheral vein);
* Mono microbial infection caused by coagulase-negative staphylococci, Enterobacteriaceae or Pseudomonas aeruginosa;
* Bacterial strain is susceptible toward gentamicin;
* Life expectancy ≥ 3 months;
* Physician in charge of the patient agrees to perform a conservative treatment;
* Calculated creatinine clearance ≥ 30 mL/min;
* Patient's informed and written consent is collected.
* For women of reproductive age: available beta-HCG dosage (with negative result) < 72h.

Non-inclusion criteria:

A patient should not be included if he presents any of the following criteria:

* Presence of any systemic complication (sepsis or septic shock, as defined by the sepsis-3 guidelines), or local complications (tunnel or port-pocket infection, thrombophlebitis, endocarditis, bone and joint infections related to the LTIVC-related BSI);
* Allergy toward aminoglycosides
* PICC-line or hemodialysis tunnelled catheter; LTIVC removal is planned within the following 3 months or LTIVC is not required for the management of the patient's underlying medical condition anymore;
* Diagnosis of LTIVC-related bloodstream infection has been made more than 3 days ago (e.g. >72 hours between the day the first blood culture drawn from the LTIVC is positive and screening visit);
* Systemic treatment of LTIVC-related bloodstream infection includes aminoglycosides (defined as a recent (<36 hours before screening visit) or ongoing systemic injection of aminoglycosides);
* Low blood ionized calcium level (<1,15 μmol/L) before injecting the first dose of genta-EDTA-Na2 lock;
* Presence of prosthetic heart valve, pacemaker or implantable defibrillator;
* The LTIVC has been inserted less than 14 days ago;
* Available Count blood cells < 72h with severe neutropenia (<500 polymorphonuclear cells/mm3);
* Subject with infection caused by Staphylococcus Aureus orCandida-spp;
* The patient is not expected to remain in hospital for at least 7 days after inclusion.
* The administration of the lock according to the protocol (24 hours/day for 48 hours and then at least 12 hours/24 hours for 5 to 8 days) is not possible.
* Decision by the referring physician to prescribe a preventive lock following curative Gentamicin-EDTA treatment (secondary prevention), between the end of treatment (D6/D9) and the D40 follow-up visit.
* Previous inclusion in a study or another therapeutic protocol requiring continuous use of the catheter
* Pregnant and breastfeeding woman;
* Protected adult subject.
* Inability to perform a blood peripheral venous sampling

Exclusion criteria

A patient should be excluded if he presents any of the following criteria:

* Presence of local or systemic complication seen on venous ultrasound performed between D2 and D5 or transthoracic echocardiography performed between Day 2 and Day 7 (D2-D7);
* GFR < 30 ml/min (between D0 and D6/9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The clinical efficacy is assessed by the frequency of clinical and microbial cure after 30 days of follow-up after the end of treatment (D40) | 30 days of follow-up after the end of treatment (D40)
  Resolution of clinical signs at the end of treatment (D6 if the patient already received 72h of a previous active lock before inclusion or D9 if he received a complete 10-day course of genta-EDTA-Na2 locks) and 30 days after completion of therapy (D40)

SECONDARY OUTCOMES:
The long-term clinical efficacy is assessed by the frequency of microbial cure after 90 days of follow-up after the end of treatment. | after 90 days of follow-up after the end of treatment (D100)
  Absence of microbial relapse (BSI with the same microbial pathogen, i.e. same species and same antibiotic susceptibility pattern) between D6-D9 and D100;

CONTACTS AND LOCATIONS:
Overall Officials: David Lebeaux, Principal Investigator — Hôpital Européen Georges Pompidou AP-HP
Locations (6):
- France (6):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - HEGP, Paris
  - Hôpital Henri Mondor, Paris
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hôpital Cochin, Paris, Île-de-France Region
  - Hôpital Beaujon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided